CLINICAL TRIAL: NCT03878680
Title: Prevalence of Asthma and Allergies Among Children in UAE-A Cross-sectional Study
Brief Title: Prevalence of Asthma and Allergies Among Children in UAE
Acronym: ISAAC-UAE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00142
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- 13-14 years age group: Children with age 13-14 years at the time of questionnaires completion, and residing in Dubai and the Northern Emirates of UAE.
  Interventions: Other: Study questionnaires
- 6-7 years age goup: Children with age 6-7 years at the time of questionnaires completion, and residing in Dubai and the Northern Emirates of UAE.
  Interventions: Other: Study questionnaires

INTERVENTIONS:
Other: Study questionnaires — Completion of the International study of Asthma and Allergies in Children(ISAAC)core questionnaires:
  1. Core questionnaire on wheezing.
  2. Core questionnaire on rhinitis.
  3. Core questionnaire on atopic dermatitis.

SUMMARY:
Multicenter, cross-sectional study to recruit a random sample of 6000 children via school class registers: 3000 children aged 13-14 years and 3000 children aged 6-7 years.

DETAILED DESCRIPTION:
Multicenter, cross-sectional study to recruit a random sample of 6000 children via school class registers: 3000 children aged 13-14 years and 3000 children aged 6-7 years.Standard ISAAC core questions for wheezing, rhinitis, and atopic dermatitis will be used. The ISAAC questionnaire has been validated by the World Health Organization and translated into many languages, and used in many countries. In this study, the Arabic and English version will be used. In addition, questions regarding exposure to Arabian incense "Bokhor" and smoking questions of the environmental questionnaire will be included.

ISAAC Questionnaires

1. Core questionnaire on wheezing.
2. Core questionnaire on rhinitis.
3. Core questionnaire on atopic dermatitis.
4. Smoking questions of the environmental questionnaire.
5. Video questionnaire on wheezing (only for 13-14 years age group, if applicable)

ELIGIBILITY:
Inclusion Criteria:

* Children with age 6 to 7 years or with age 13 to 14 years at the time of questionnaires completion, and residing in Dubai and the Northern Emirates of UAE.
* Children aged 6 to 7 years or 13 to14 years, whose legal guardians give their consent.
* Able to give assent in the 13 to 14 years group.
* Able to comprehend and answer the questionnaire themselves in the 13 to 14 years group.

Exclusion Criteria:

* Aged 13 to 14 years and unable to answer the questionnaire due to physical or mental disability.
* Parent or legal guardian refuses sign and return consent for the 6 to 7 years group and the 13 to 14 years group.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with age 6-7 years or with age 13-14 years at the time of questionnaires completion, and residing in Dubai and the Northern Emirates of UAE
Sampling Method: Probability Sample
Enrollment: 3737 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Prevalence of asthma in children aged 6-7 years and 13-14 years in Dubai and the Northern Emirates. | 3 Month
  Through International study of Asthma and Allergies in Children(ISAAC)core questionnaire on Asthma and Wheezing: A set of 8 questions to address wheezing attacks, assessing the prevalence of wheezing illness, frequency of wheezing, diagnosis of asthma.Descriptive summaries of the data will be presented. Comparisons between different centers on the rates of events will be made using appropriate methods. Crude rates can be compared by using contingency tables or logistic regression. Comparison of standardized rates or data that needs controlling for confounding will require analysis by logistic regression

SECONDARY OUTCOMES:
Severity of asthma in children aged 6-7 years and 13-14 years in Dubai and the Northern Emirates. | 3 Month
  Through International study of Asthma and Allergies in Children(ISAAC)core questionnaire on (a)Wheezing,(b)rhinitis and (c)atopic dermatitis.
  1. Wheezing questionnaire:8 questions to address wheezing attacks, frequency, assessing prevalence illness, diagnosis of asthma.
  2. Rhinitis questionnaire : 6 questions to addressing detection of rhinitis, detecting atopy among subjects with rhinitis , interference with daily activities.
  3. Atopic Dermatitis questionnaire : 7 questions to addressing severity, rashes, and nonatopic forms of eczema.
     * Most of the questions used iare Binary questions Yes or NO .
     * Data from 6-7 year old and 13-14 year old analysis separately. Each measure of prevalence and severity will be compared between centres. The effect of cluster sampling by schools will considered in the analysis.
     * Basic descriptive summaries data will be compiled and presented for each condition, in both age groups, for males and females, from each centres.

OTHER OUTCOMES:
Prevalence of asthma in children aged 6-7 years and 13-14 years in Dubai and the Northern Emirates, who were exposed to Arabian incense "Bokhor". | 3 Month
  Questionnaire of Exposer to Arabian incense "Bokhor"
Prevalence of asthma in children aged 6-7 years and 13-14 years in Dubai and the Northern Emirates, who were exposed to tobacco smoke | 3 Month
  Smoking questions of the environmental questionnaire

CONTACTS AND LOCATIONS:
Locations (6):
- United Arab Emirates (6):
  - Research Site, Ajman
  - Research Site, Dubai
  - Research Site, FUJ
  - Research Site, Ras al-Khaimah
  - Research Site, Sharjah city
  - Research Site, UMQ

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2287R00142&attachmentIdentifier=170b8f20-7342-4be5-8be3-1418920f8b17&fileName=4.0_ISAAC_D2287R00142_CSR_final_V1.0_(08Apr2020)_Docusign_Redacted_for_CT.Gov.pdf&versionIdentifier=